CLINICAL TRIAL: NCT04910776
Title: An Open-label, Multinational, Multicenter, Intravenous Infusion Study of the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Avalglucosidase Alfa in Treatment naïve Pediatric Participants With Infantile-Onset Pompe Disease (IOPD)
Brief Title: Clinical Study for Treatment-naïve IOPD Babies to Evaluate Efficacy and Safety of ERT With Avalglucosidase Alfa
Acronym: Baby-COMET
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC14462; U1111-1246-6645 (Registry Identifier: ICTRP); 2024-513859-33 (Registry Identifier: CTIS); 2020-004686-39 (EudraCT Number)
Record Dates: First submitted 2021-05-25; First posted 2021-06-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Glycogen Storage Disease Type II
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avalglucosidase alfa (Experimental): Administered intravenously every 2 weeks
  Interventions: Drug: avalglucosidase alfa

INTERVENTIONS:
Drug: avalglucosidase alfa — Sterile lyophilized powder intravenous (IV) infusion
  Other Names: GZ402666

SUMMARY:
This is a single group, treatment, Phase 3, open-label study to assess efficacy, safety, pharmacokinetic (PK), pharmacodynamics (PD) of avalglucosidase alfa in treatment-naïve male and female participants with IOPD.

Study details include:

* Study duration: Screening - up to 4 weeks;
* Primary Analysis Period (PAP) - 52 weeks;
* Extended Treatment Period (ETP) - 52 weeks;
* Extended Long term Treatment Period (ELTP) - 104 weeks; 4-week follow-up period for a total study duration - up to 4.08 years.
* Treatment duration: Up to 4 years
* Visit frequency: every other week and potentially every week

DETAILED DESCRIPTION:
Study duration may be variable by country, including at least completion of the PAP and ETP, and up to 4.08 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have confirmed diagnosis of infantile-onset Pompe disease defined as: the presence of 2 lysosomal acid α-glucosidase (GAA) pathogenic variants and a documented GAA deficiency from blood, skin, or muscle tissue; or the presence of 1 GAA pathogenic variant and a documented GAA deficiency from blood, skin and muscle tissue in 2 separate samples (from either 2 different tissues or from the same tissue but at 2 different sampling dates).
* Participants must have established cross-reactive immunological material (CRIM) status available prior to enrollment.
* Participants must have cardiomyopathy at the time of diagnosis: ie, left ventricular mass index (LVMI) equivalent to mean age specific LVMI

  * +1 standard deviation for participants diagnosed by newborn screening or sibling screening;
  * +2 standard deviation for participants diagnosed by clinical evaluation.
* Parents or legally authorized representative(s) must be capable of giving signed informed consent.

Exclusion Criteria:

* Participants with symptoms of respiratory insufficiency, including any ventilation use (invasive or noninvasive) at the time of enrollment.
* Participants with major congenital abnormality.
* Participants with clinically significant organic disease (with the exception of symptoms relating to Pompe disease).
* Participant received any Pompe disease specific treatment, eg enzyme-replacement gene therapy (ERT).
* Participant who has previously been treated in any clinical trial of avalglucosidase alfa.
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 0 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-03-06 (Estimated); Study Completion 2027-08-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who are alive and free of invasive ventilation at Week 52 | Week 52

SECONDARY OUTCOMES:
Proportion of participants who are alive and free of invasive ventilation at 12 and 18 months of age | at 12 and 18 months of age
Proportion of participants who are alive at Week 52 | Week 52
Proportion of participants who are alive at 12 and 18 months of age | at 12 and 18 months of age
Proportion of participants who are free of ventilator use (invasive and non-invasive separate and combined) at Week 52 | Week 52
Proportion of participants who are free of supplemental oxygen use at Week 52 | Week 52
Change from baseline to Week 52 in left ventricular mass (LVM)-Z score | Week 52
Change from baseline to Week 52 in Alberta Infant Motor Scale (AIMS) score | Week 52
Change from baseline to Week 52 in body length Z-scores | Week 52
Change from baseline to Week 52 in body weight Z-scores | Week 52
Change from baseline to Week 52 in head circumference Z-scores | Week 52
Change from baseline to Week 52 in body length percentiles | Week 52
Change from baseline to Week 52 in body weight percentiles | Week 52
Change from baseline to Week 52 in head circumference percentiles | Week 52
Change from baseline to Week 52 in urinary Hex4 | Week 52
Number of participants experiencing at least 1 treatment-emergent adverse events (TEAE), including infusion associated reactions (IAR) | Week 52, Week 212
Number of participants with abnormalities in physical examinations | Week 52, Week 208
Number of participants with potentially clinically significant abnormality (PCSA) in clinical laboratory results | Week 52, Week 208
Number of participants with PCSA in vital signs measurements | Week 52, Week 208
Number of participants with PCSA in 12-lead electrocardiogram (ECG) | Week 52, Week 208
Incidence of treatment-emergent anti-drug antibodies (ADA) | Week 52, Week 208
Plasma concentration of avalglucosidase alfa | at Day 1, Week 12, and Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- United States (6):
  - Stanford Hospital- Site Number : 8400006, Stanford, California
  - Children's Hospitals and Clinics of Minnesota- Site Number : 8400008, Minneapolis, Minnesota
  - Advanced Medical Genetics- Site Number : 8400002, Hawthorne, New York
  - Duke University Medical Center- Site Number : 8400004, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center- Site Number : 8400001, Cincinnati, Ohio
  - Seattle Children's Hospital- Site Number : 8400003, Seattle, Washington
- Investigational Site Number : 0560001, Leuven, Belgium
- China (2):
  - Investigational Site Number : 1560002, Qingdao
  - Investigational Site Number : 1560001, Shanghai
- Investigational Site Number : 2760001, Bad Oeynhausen, Germany
- Investigational Site Number : 3800002, Monza, Lombardy, Italy
- Investigational Site Number : 5280001, Rotterdam, Netherlands
- Investigational Site Number : 7240001, Esplugues de Llobregat, Catalunya [Cataluña], Spain
- Investigational Site Number : 1580001, Taipei, Taiwan
- United Kingdom (2):
  - Investigational Site Number : 8260001, London, London, City of
  - Investigational Site Number : 8260002, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org